CLINICAL TRIAL: NCT04284761
Title: A Study to Establish the Feasibility of Biolen for the Local Delivery of Bicalutamide in Patients With Prostate Cancer
Acronym: Biolen-PC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alessa Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-001
Record Dates: First submitted 2020-02-12; First posted 2020-02-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-08

CONDITIONS: Prostate Adenocarcinoma; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — bicalutamide

STUDY DESIGN:
Intervention Model Description: Biolen bicalutamide implant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Biolen (Experimental): Biolen bicalutamide implant. Single implantation. In situ until prostatectomy
  Interventions: Combination Product: Bicalutamide implant

INTERVENTIONS:
Combination Product: Bicalutamide implant — Biolen bicalutamide implant

SUMMARY:
Biolen, a novel implant, is intended to deliver an anti-androgen locally to the prostate gland for the management of prostate disease, while minimizing systemic exposure and its associated side-effects. The objectives of the study are to assess whether the Biolen is safe.

DETAILED DESCRIPTION:
This prospective, multi-center, single-arm feasibility study is planned to assess the safety and patient tolerance of Biolen for the localized delivery of bicalutamide into the prostate in patients presenting for treatment of prostate cancer. Study participants will have placement of the drug eluting Biolen and be followed through scheduled radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Study participant qualified and planning for radical prostatectomy.
* At least 1 prostate lesion measurable by MRI > 0.5 cm within one month of screening.
* PSA > 3 ng/mL within 3 months of screening.
* Gleason score 3+4 or higher.
* Study participant must be willing to undergo post-treatment imaging by MRI.
* ECOG performance status 0 or 1.

Exclusion Criteria:

* Prior radiotherapy or surgery for prostate cancer.
* Prior or ongoing hormonal therapy for prostate cancer.
* Prior prostate procedures such as transurethral resection of the prostate, transurethral microwave thermotherapy of the prostate, high-intensity focused ultrasound or minimally invasive BPH procedure.
* Study participant unwilling or unable to undergo MRI, including patients with contra-indications to MRI, such as cardiac pacemakers, non-compatible intracranial vascular clips, etc.
* Metallic hip implant or any other metallic implant or device that distorts the quality of prostatic MR images.
* Use of 5 alpha reductase inhibitors (e.g. Finasteride or Dutasteride) within 3 months of screening or total use within the last two years prior to screening of > 3 months.
* Presence of any metastatic disease.
* Prostate volume more than 80 cc at prior MRI imaging.
* I-PSS score >20.
* History of prostate infection.

Min Age: 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Safety as measured by number and incidence of adverse events | change from baseline to radical prostatectomy up to 12 weeks after implantation
  Adverse Events

SECONDARY OUTCOMES:
change in prostate size | change from baseline to radical prostatectomy up to 12 weeks after implantation
  prostate measurement by MRI
change in tumor size | change from baseline to radical prostatectomy up to 12 weeks after implantation
  tumor measurement by MRI
change in Prostate Specific Antigen (PSA) | change from baseline to radical prostatectomy up to 12 weeks after implantation
  PSA level

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Munster, MD, Study Director — Alessa Therapeutics Inc.
Locations (4):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Australia (2):
  - Australian Clinical Trials, Wahroonga, New South Wales
  - University of Wollongong, Wollongong, New South Wales
- Tauranga Urology Research, Tauranga, North Island, New Zealand

IPD SHARING:
Plan to Share IPD: No